CLINICAL TRIAL: NCT07156487
Title: The Evaluation of the Effects of Computer-controlled Electronic Anesthesia Systems and Traditional Local Anesthesia Techniques, Along With Different Anesthetic Agents, on Pain and Anxiety Levels During Dental Treatments in Pediatric Patients: A Randomized Controlled Clinical Study
Brief Title: Pain and Anxiety in Pediatric Dentistry: Computer-Controlled vs. Traditional Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dicle University (Other)
Responsible Party: Principal Investigator, Hasan Said Şener, Research Asisstant, Dicle University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HRÜ/25.06.54
Record Dates: First submitted 2025-05-01; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Traditional Local Anesthesia; Computer-controlled Electronic Anesthesia; Dental Anxiety; Anxiety in Children
Keywords: Pediatric Dentistry; Injections, Intraosseous; Dental Instruments
MeSH Terms: interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: The study was a single-center randomized controlled trial using a split mouth design
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Dental Anesthesia (CCLAD - Computer Controlled Local Anesthetic Delivery) (Experimental): For Maxillary Teeth: For maxillary teeth, the SleeperOne® 5 electronic local anesthesia system was used. After confirming pulp vitality through a cold or electric pulp test, the target area was dried, and 10% lidocaine topical anesthetic was applied for 1 minute using a cotton pellet. Then, 1.7 ml of Ultracaine D-S Fort was delivered via intraosseous injection using a 30-gauge, 9 mm Effitec needle in pediatric mode.
  For Mandibular Teeth: For mandibular teeth, the SleeperOne® 5 electronic local anesthesia system was used to perform intraosseous injection in pediatric mode. Prior to the injection, pulp vitality was assessed using a cold or electric pulp test. The injection site was then dried, and 10% lidocaine topical anesthetic spray was applied with a cotton pellet for 1 minute. Following this, 1.7 ml of Ultracaine D-S Fort was administered using a 30-gauge, 9 mm Effitec needle.
  Interventions: Device: Digital Anesthesia with SleeperOne 5
- Traditional Local anesthesia Techniques (Active Comparator): For the contralateral maxillary teeth:
  After confirming vitality, the site is dried and 10% lidocaine spray is applied for 1 minute. Buccal infiltration is performed. The cheek and lip are retracted, mucosa tightened, and the needle inserted at the tooth apex. After bone contact, the needle is withdrawn 1 mm, aspirated, and Ultracaine D-S Fort injected slowly over 1 minute using a 30G, 16 mm Effitec needle and metal carpule syringe.
  For the contralateral mandibular teeth:
  The retromolar area is dried, and 10% lidocaine spray is applied with a cotton pellet for 1 minute. After retracting the cheek and lip, the needle is inserted between the pterygomandibular raphe and internal oblique ridge, aligned with the contralateral molars. After bone contact, aspiration is performed. Ultracaine D-S Fort is slowly injected over 1 minute using a traditional metal carpule syringe and a 27-gauge, 35 mm Effitec needle following the standard inferior alveolar nerve block technique.
  Interventions: Device: Infiltration Anesthesia with a Metal Cartridge Syringe; Device: Mandibular Block Anesthesia with a Metal Cartridge Syringe

INTERVENTIONS:
Device: Digital Anesthesia with SleeperOne 5 — For both maxillary and mandibular teeth, 1.7 mL of Ultracaine D-S Fort carpule (4% articaine with 1:200,000 epinephrine) was administered in two stages (gingival and intraosseous injection) using a computer-controlled intraosseous anesthesia system with a 30-gauge, 9 mm Effitec needle.
  Other Names: SleeperOne 5
  Arms: Digital Dental Anesthesia (CCLAD - Computer Controlled Local Anesthetic Delivery)
Device: Infiltration Anesthesia with a Metal Cartridge Syringe — For maxillary teeth, buccal infiltration is performed using a metal carpule syringe and a 30G, 16 mm Effitec needle (Dental Hi Tec, France); after aspiration, Ultracaine D-S Fort is slowly injected over 1 minute.
  Other Names: Supraperiosteal Anesthesia
  Arms: Traditional Local anesthesia Techniques
Device: Mandibular Block Anesthesia with a Metal Cartridge Syringe — For mandibular teeth, the injection site is dried, and a 27G, 35 mm Effitec needle (Dental Hi Tec, France) is inserted between the pterygomandibular raphe and internal oblique ridge, aligned with contralateral molars. After aspiration, Ultracaine D-S Fort is slowly injected over 1 minute using a traditional metal carpule syringe, following the standard mandibular block technique.
  Other Names: IANB
  Arms: Traditional Local anesthesia Techniques

SUMMARY:
The purpose of this clinical study is to evaluate how different local anesthesia techniques affect pain and anxiety levels in children undergoing dental treatment. Specifically, the study compares traditional syringe-based anesthesia with a computer-controlled local anesthesia system.

The study seeks to answer the following question: Which combination of anesthesia technique is most effective in reducing pain and anxiety in pediatric dental patients?

By understanding the impact of these variables, the study aims to help dental professionals choose the most appropriate anesthesia approach to improve the comfort and emotional well-being of children during dental procedures.

DETAILED DESCRIPTION:
This randomized controlled clinical trial will be conducted at the Department of Pediatric Dentistry, Faculty of Dentistry, Dicle University. The study will include 84 voluntary pediatric patients aged between 7 and 10 years who meet the eligibility criteria defined.These patients will be selected among those who present with a clinical need for pulpotomy or pulpectomy proce dures in their primary molar teeth located in either the upper or lower jaws. Prior to any intervention, patients and their legal guardians will be fully informed about the study, and written informed consent will be obtained. The study aims to evaluate and compare the impact of traditional local anesthesia techniques and computer-controlled local anesthetic delivery systems (CCLAD) on children's pain and anxiety levels during dental procedures.

In a within-subject crossover design, both traditional (syringe-based) and computer-controlled anesthesia methods will be applied to the same patient but on different sides of the mouth. This design enables objective comparisons and minimizes inter-individual variability. A total of 42 patients will be included in each group, with each child serving as their own control. Local anesthesia will be administered to teeth requiring treatment either on the left or right side, depending on the clinical indication.

The primary and secondary outcome measures will include assessments of both physiological and psychological parameters. Pain and anxiety will be measured using a combination of psychometric, physiological, and biochemical evaluation methods. These include:

Physiological measurements: heart rate, oxygen saturation (SpO₂) and body temperature.

Psychometric scales:

Facial Image Scale (FIS) Visual Analog Scale (VAS) Wong-Baker Faces Pain Rating Scale (WBS) Modified Child Dental Anxiety Scale (MCDAS) Children's Fear Survey Schedule-Dental Subscale (CFSS-DS) FLACC Behavioral Pain Scale (Face, Legs, Activity, Cry, Consolability) Data from these assessments will be recorded for both groups and analyzed to determine which anesthesia technique provides the best outcome in terms of minimizing pain and anxiety.

Although this is not a patient registry study, quality assurance measures will be applied to ensure data integrity. These include:

Regular validation checks for consistency and completeness during data entry. Source data verification against patient records and clinical forms. A standardized data dictionary defining all variables used, including their measurement units and coding schemes where applicable.

Implementation of standard operating procedures (SOPs) for participant enrollment, data collection, safety monitoring, and data management.

Statistical analyses will be planned according to a predefined protocol, using appropriate tests to evaluate differences between interventions.

A sample size calculation has been performed to ensure that 84 patients are sufficient to detect clinically significant differences.

A missing data management plan is in place to handle incomplete or inconsistent entries, ensuring statistical robustness and data quality.

This study is expected to contribute valuable evidence to the field of pediatric dentistry by identifying the most effective and child-friendly local anesthesia method, thereby improving patient care and treatment experiences.

ELIGIBILITY:
Inclusion Criteria:

* Patients classified as ASA I in general systemic health

  * Children between 7 and 10 years of age
  * Absence of any syndromic condition
  * No physical or mental disability
  * No prior dental treatment experience
  * Frankl Behavior Rating Scale Class III or IV
  * Presence of carious lesions limited to less than one-third of the buccolingual distance between cusp tips on the occlusal surfaces of primary or permanent molars on both sides
  * Radiographic evidence of caries involving up to half of the dentin thickness with intact dentin at the pulp-dentin border in primary or permanent molars on both sides
  * Teeth on both sides responding positively to pulp vitality tests, with no periradicular pathology or significant widening of the lamina dura on periapical radiographs

Exclusion Criteria:

* Patients with mild or severe systemic diseases or those undergoing medical treatment

  * Patients younger than 7 or older than 10 years of age
  * Uncooperative or noncompliant patients classified as Class I or Class II according to the Frankl Behavior Rating Scale
  * Patients requiring urgent dental treatment
  * Patients with wide carious lesions extending beyond one-third of the buccolingual distance between cusp tips on the occlusal surfaces
  * Patients with carious lesions limited to less than one-third of the buccolingual width only on one side of the jaw
  * Teeth with carious lesions not reaching half of the dentin thickness on radiographic evaluation or lacking intact dentin at the pulp border
  * Teeth that do not respond positively to pulp vitality tests, or that show periradicular lesions or marked widening of the lamina dura on periapical radiographs

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To assess the patient's pain level (Before and after anesthesia) | through study completion, an average of 6 month.
  Wong-Baker Faces Pain Rating Scale The scale contains a series of six faces ranging from a happy face at 0 to indicate "no hurt" to a crying face at 10 to indicate "hurts worst".
To assess the patient's pain level (During anesthesia) | through study completion, an average of 6 month.
  The Visual Analog Scale (VAS) is a unidimensional tool used to measure pain intensity on a continuous spectrum, ranging from "no pain" to "worst imaginable pain." It consists of a 10 cm line with descriptive anchors at both ends. In our study, VAS will be applied as a 10 cm horizontal line marked at 1 cm intervals to quantify pain levels.
To assess the patient's pain level (During anesthesia) | through study completion, an average of 6 month.
  Behavioral responses were recorded using the FLACC scale, which evaluates Face, Legs, Activity, Cry, and Consolability. Each domain is scored from 0-2, for a total range of 0-10.
To assess the patient's anxiety level (Before anesthesia ) | through study completion, an average of 6 month.
  The CFSS-DS is a validated psychometric scale developed in 1982 to assess dental anxiety in children. It includes items scored from 1 (not afraid) to 5 (very afraid). Total scores indicate anxiety levels as follows:
  <38: No anxiety
  38-45: Moderate dental anxiety
  >45: Severe dental anxiety
To assess the patient's anxiety level (Before and after anesthesia) | through study completion, an average of 6 month.
  Facial Image Scale (FIS) The Facial Image Scale (FIS) is a projective tool designed to quickly assess pre-procedural anxiety levels in young children, starting from age 3. It consists of five faces, ranging from very happy (score = 1) to very unhappy (score = 5), reflecting increasing levels of fear.
Pulse rate measurement to assess patient's dental anxiety (Before,after and during anesthesia) | through study completion, an average of 6 month.
  Measurement will be made with a pulse oximeter.The measurement will be performed using a pulse oximeter attached to the patient's fingertip.
Blood oxygen saturation measurement to assess patient's dental anxiety (Before,after and during anesthesia) | through study completion, an average of 6 month.
  Measurement will be made with a pulse oximeter.The measurement will be performed using a pulse oximeter attached to the patient's fingertip.
Body temperature measurement to assess the patient's anxiety (Before,after and during anesthesia) | through study completion, an average of 6 month.
  Tympanic Temperature Measurement
  Under stress or anxiety, adrenaline increases heart rate and body temperature. Tympanic thermometers measure core temperature through the tympanic membrane, providing accurate, non-invasive, and rapid readings. This method is effective in ICU settings for both adults and children, offering advantages like minimal infection risk and resistance to environmental changes.

SECONDARY OUTCOMES:
Pulse rate measurement to assess opetator's anxiety (Before,after and during anesthesia) | through study completion, an average of 6 month.
  The measurement will be performed using a pulse oximeter attached to the operator's fingertip.
Body temperature measurement to assess the operator's anxiety (Before,after and during anesthesia) | through study completion, an average of 6 month.
  Tympanic Temperature Measurement Under stress or anxiety, adrenaline increases heart rate and body temperature. Tympanic thermometers measure core temperature through the tympanic membrane, providing accurate, non-invasive, and rapid readings. This method is effective in ICU settings for both adults and children, offering advantages like minimal infection risk and resistance to environmental changes.
Blood oxygen saturation measurement to assess operator's anxiety (Before,after and during anesthesia) | through study completion, an average of 6 month.
  The measurement will be performed using a pulse oximeter attached to the operator's fingertip

CONTACTS AND LOCATIONS:
Overall Officials: Emin C Tümen, Study Director — Dicle Universty
Locations (1):
- Dicle University Faculty of Dentistry, Department of Pediatric Dentistry, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 months after publication of results
Access Criteria: dentists, medicine doctors

REFERENCES:
- See also: VAS (Visual Analog Scala): — https://www.spinetr.com/uploads/files/skor/vizuelanalogskala.pdf
- See also: WBS (Wong-Baker Facesl Pain Rating Scale) — https://wongbakerfaces.org/wp-content/uploads/2016/11/FACES_Publication_Turkish_Black_w-instructions.pdf
- See also: flacc scale — https://www.mdcalc.com/calc/10545/face-legs-activity-cry-consolability-flacc-scale?utm

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-07-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT07156487/Prot_SAP_ICF_000.pdf